CLINICAL TRIAL: NCT03475173
Title: New Non-invasive Modalities for Assessing Retinal Structure and Function:Preliminary Investigation
Brief Title: New Non-invasive Modalities for Assessing Retinal Structure and Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Randy Kardon (Other)
Responsible Party: Sponsor-Investigator, Randy Kardon, Dr. Randy Kardon M.D. Ph.D Professor and Director of Neuro-ophthalmology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201611825
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Optic Neuropathy; Branch Retinal Artery Occlusion; Hemianopia; Leber Hereditary Optic Neuropathy; Acute Zonal Occult Outer Retinopathy
Keywords: Optic Neuropathy; , Retinopathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic; Retinal Artery Occlusion; Hemianopsia; Optic Atrophy, Hereditary, Leber; Acute zonal occult outer retinopathy; Optic Nerve Diseases; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laser Speckle Blood Flow Group (Experimental)
  Interventions: Device: LSFG-NAVI

INTERVENTIONS:
Device: LSFG-NAVI — laser-speckle blood flow of ocular arteries and veins

SUMMARY:
This study investigates a new technology to assess the structure and function inside the eye. Retinal imaging of subjects with inner and outer retinal defects to detect areas of abnormal structure and function compared to other visual function tests.

ELIGIBILITY:
Controls:

Inclusion:

Normal eye exam in last 2 years

Exclusion:

Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay. Any abnormalities of the retina or optic nerve that could affect metabolism of the retina outside of normal.

Subjects with Inner Retina Defect:

Inclusion:

Defined structural defect to include those with Ischemic optic neuropathy, branch retinal artery occlusion (BRAO), hemianopia or visual field defect that respects the vertical meridian, inherited mitochondrial optic neuropathies such as Leber's and Dominant Optic Neuropathy, other retinopathies or optic neuropathies.

Exclusion:

Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.

Subjects with Outer Retinal Defect:

Inclusion:

AZOOR (acute zonal occult outer retinopathy) or other focal or diffuse outer photoreceptor loss of function

Exclusion:

Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.

The 450 total is to allow for exclusion of some subjects or in the event that the enrolled subject blinks too much or cannot fixate on a visual target adequately to maintain the same eye position during the short imaging interval. We hope to have a total of 450 (50 controls and 400 patients)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Ocular Blood Flow | 1 day
  imaging the movement of blood through blood vessels in retina and optic nerve

CONTACTS AND LOCATIONS:
Overall Officials: Randy H Kardon, MD, PhD, Principal Investigator — University of Iowa Department of Ophthalmology
Locations (1):
- University of Iowa Department of Ophthalmology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No